CLINICAL TRIAL: NCT05270174
Title: A Prospective, Multicenter Cohort Study of Urinary Exosome lncRNAs for Preoperative Diagnosis of Lymphatic Metastasis in Patients With Bladder Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: SYSEC-KY-KS-2021-278
Record Dates: First submitted 2022-02-09; First posted 2022-03-08 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2022-02

CONDITIONS: Explore Whether lncRNA-ElNAT1 in Urine Exosomes Can be Used as a New Target for Preoperative Diagnosis of Lymph Node Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- lncRNA-ELNAT1 high expression group
  Interventions: Other: no intervention
- lncRNA-ELNAT1 low expression group
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
Bladder cancer is one of the most frequent malignant tumors of the urinary system in China, seriously threatening the life safety of patients. The main treatment methods for bladder cancer include surgical resection, radiotherapy and chemotherapy, immunotherapy, and targeted therapy, among which surgical resection is still the only reliable radical treatment at present. Lymphatic metastasis is the main mode of metastasis of bladder cancer, and preoperative diagnosis is of great significance to determine whether radical surgical treatment can be performed for some patients with advanced bladder cancer. Recent studies reveal that exosomes, as key signaling molecules in the tumor microenvironment, have been confirmed to be associated with various tumor progressions. Our previous study showed that lncRNA-ELNAT1 highly expressed in urine exosomes of bladder cancer patients can promote lymphatic metastasis of bladder cancer by inducing lymphatic angiogenesis, and is associated with poor prognosis of patients. However, whether exosome ELNAT1 can be used as an independent preoperative predictor of lymph node metastasis of bladder cancer needs to be explored in further clinical trials, and this study will further clarify the association between the two. In this study, urine exosomes were collected from positive and negative control patients with lymph node metastasis of bladder cancer, and the ROC curve was statistically analyzed and fitted to determine whether exosome ELANT1 could be used as an independent predictor of lymph node metastasis of bladder cancer.

DETAILED DESCRIPTION:
1. According to the selection criteria. Bladder cancer patients with informed consent in the study were first included.
2. The patients with indications of radical cystectomy were selected.
3. Urine samples were collected before radical cystectomy and exocrine bodies were extracted to analyze the expression level of ELNAT1
4. According to the postoperative lymph node pathological results, the above patients were further divided into two groups：lymphatic metastasis positive group and negative group.
5. We perform statistical analysis of urinary exosomal ELNAT1 to validate the performance of diagnosing lymphatic metastasis of bladder cancer

ELIGIBILITY:
Inclusion Criteria:

1. Patients older than 18 years old
2. Clinically diagnosed urothelial carcinoma bladder cancer
3. Patients agreed to provide the urine sample
4. Patients who voluntarily agreed to informed consent

Exclusion Criteria:

1. Patients with distant metastasis
2. Patients with uncontrolled viral infection (HIV, HBV, HCV)
3. Patients who are pregnant, or have the possibility of pregnancy and are on lactating
4. Hypersensitivity or history of allergic to the drug being used
5. Patients with cerebrovascular disease, complications, and infections that are not medically controlled
6. Patients with a history of other malignant diseases within the past 5 years (excluding cured non-melanoma skin cancer or in situ cervical cancer)
7. Those who are taking drugs that can cause drug interactions with chemotherapy
8. Patients who withdraw consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the patient diagnosed with bladder cancer
Sampling Method: Probability Sample
Enrollment: 74 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Lymph node metastases in bladder cancer | 1 years
  Analyses of number and location of lymph node metastases based on pathological diagnosis

SECONDARY OUTCOMES:
recurernce rate | 3 years
  The rate of recurrence will be detected after radical cystectomy by postoperative follow-up visit

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen Memorial Hosptial, Guangzhou, China